CLINICAL TRIAL: NCT07050706
Title: Study on the Correlation Between Serum PRMT5 Level and Cardiac Structural and Functional Indicators in Patients With Heart Failure
Brief Title: The Correlation Between Serum PRMT5 Level and Cardiac Ultrasound Indicators in Patients With Heart Failure
Status: Enrolling by invitation | Type: Observational
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Cai Sidong, assistant research fellow, The University of Hong Kong-Shenzhen Hospital
Other Study IDs: PRMT5 and Heart Failure; 82300446 (Other Grant/Funding Number: National Science Foundation of China); 2022A1515111093 (Other Grant/Funding Number: Guangdong Basic and Applied Basic Research Foundation); RCBS20231211090745071 (Other Grant/Funding Number: Shenzhen Science and Technology Program)
Record Dates: First submitted 2025-06-13; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure, Systolic
Keywords: PRMT5; Heart failure; cardiac function and cardiac structure
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pathological cardiac hypertrophy is characterized by abnormal cardiomyocyte metabolism, reduced myocardial contractility, and dysregulated synthesis of myocardial contractile proteins. This pathological process leads to progressive impairment of cardiac function and ultimately progresses to heart failure. Previous studies have demonstrated that PRMT5 exerts a significant inhibitory effect on heart failure, yet its clinical significance in the context of heart failure remains undefined. In this study, we hypothesized that serum PRMT5 may serve as a biomarker to predict cardiac structural parameters and functional indices. Therefore, we aim to analyse the correlation between serum PRMT5 levels and the following parameters-LVPWs, LVPWd, LVIDs, LVIDd, IVSTs, IVSTd, EF, FS, LVMi and RWT on the first day when participants are enrolled in this study.

DETAILED DESCRIPTION:
The aim of this study is to collect blood samples from both healthy controls and heart failure patients and to clarify the correlation between serum PRMT5 levels on the first day of enrollment and cardiac ultrasound indicators. Serum PRMT5 levels are measured by means of enzyme-linked immunosorbent assay (ELISA). Left ventricular posterior wall thickness at end-systole (LVPWs), Left ventricular posterior wall thickness at end-diastole (LVPWd), left ventricular internal diameter at end-systole (LVIDs), left ventricular internal diameter at end-diastole (LVIDd), interventricular septum at end-systole (IVSTs) and interventricular septal septum at end-diastole (IVSTd) are measured on the first day of enrollment via echocardiography. Ejection fraction (EF), fractional shortening (FS), left ventricular mass index (LVMi), and relative wall thickness (RWT) are subsequently calculated based on LVIDd, LVPWd, and IVSTd values. Finally, the correlations between serum PRMT5 levels and the following indicators are analyzed: LVPWs, LVPWd, LVIDs, LVIDd, IVSTs, IVSTd, EF, FS, LVMi and RWT.

ELIGIBILITY:
Inclusion Criteria:

Healthy group: Aged ≥18 years (both sexes), systolic blood pressure (SBP) ≤120 mmHg and diastolic blood pressure (DBP) ≤80 mmHg, no history of cardiovascular diseases, ejection fraction (EF) ≥50%.

Heart failure group: Aged ≥18 years (both sexes), EF ≤50%.

Exclusion Criteria:

* Exclusion criteria for healthy people: people with other underlying diseases or congenital diseases are not included in the study.
* Exclusion criteria for patients with heart failure: patients with heart failure other metabolic diseases or congenital diseases were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study evaluated whether serum PRMT5 levels could predict echocardiographic parameters in healthy controls and heart failure patients. A total of 50 participants in the healthy group and 50 in the heart failure group completed the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum PRMT5 level at baseline | Baseline (day of informed consent agreement and blood sampling)
  Serum PRMT5 level is analysed at the day of informed consent agreement and blood sampling
LVIDs level at baseline | Baseline
  Left ventricular internal diameter at systolic state is measured at the day of informed consent agreement and cardiac ultrasound examination
LVIDd level at baseline | Baseline
  Left ventricular internal diameter at diastolic state is measured at the day of informed consent agreement and cardiac ultrasound examination
LVPWs level at baseline | Baseline
  left ventricular posterior wall at systolic state is measured at the day of informed consent agreement and cardiac ultrasound examination
LVPWd level at baseline | Baseline
  left ventricular posterior wall at diastole state is measured at the day of informed consent agreement and cardiac ultrasound examination
IVSTs at baseline | Baseline
  Interventricular septum at systolic state is measured at the day of informed consent agreement and cardiac ultrasound examination
IVSTd at baseline | Baseline
  Interventricular septum at diastolic state is measured at the day of informed consent agreement and cardiac ultrasound examination
EF at baseline | Baseline
  Ejection fraction is calculated according to the formula below:
  1. EF=(LVEDV-LVESV)/LVEDV*100%;
  2. LVEDV=(7.0*LVIDd^3)/(2.4+LVIDd)
  3. LVESV=(7.0*LVIDs^3)/(2.4+LVIDs)
FS at baseline | Baseline
  Fractional shortening is calculated based on the formula below:
  FS=(LVIDd-LVIDs)/LVIDd*100%
LVMi at baseline | Baseline
  Left ventricular mass index is calculated according to the formula below:
  1. LVMi(g/m^2)=LVM/BSA;
  2. LVM(g)=LVM=0.8×1.04×[(LVIDd+IVSd+LVPWd)^3-LVIDd^3]+0.6;
  3. BSA(m^2)=0.007184×W^0.425×H^0.725 (W: Weight, kg; H: Height, cm)
RWT at baseline | Baseline
  Relative wall thickness is calculated according to the formula below:
  RWT=2*(IVSd+LVPWd)/LVIDd

CONTACTS AND LOCATIONS:
Overall Officials: Assistant research fellow, Principal Investigator — The University of HongKong-Shenzhen Hospital
Locations (1):
- the University of Hongkong-Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided